CLINICAL TRIAL: NCT03635866
Title: PET/MRI Study of Men With Highly Suspicious MRI Lesions That Showed no Clinically Significant Prostate Cancer Following MRI Fusion Targeted Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-00601
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prior negative MRFTB of PI-RADS 4 and 5 lesions (Experimental): Diagnosed withing 12 months of initial diagnostic cancer biopsy
  Interventions: Diagnostic Test: Fluciclovine PET/MRI

INTERVENTIONS:
Diagnostic Test: Fluciclovine PET/MRI — It is unknown how many negative MRFTBs of PI-RADS 4 lesions are false negative biopsies or false positive tests.

SUMMARY:
The principal aim of this study is to determine if PET/MRI imaging with 18-F fluciclovine (Axumin) identifies those men with false negative MRI fusion targeted biopsy (MRFTB) of PI-RADS 4 and 5 lesions. PI-RADS 4 and 5 MRI lesions are highly suspicious for clinically significant prostate cancer and require future repeat MRI imaging and possible repeat prostate biopsy depending on the results of the repeat MRI. Men, who had negative MRFTB within past 12 months of PI- RADS 4 or 5 MRI lesion will be included in this diagnostic study. The repeat MRI is standard of care at NYU Langone Health. The investigation aspect of the study is to perform an Axumin scan the same day as the MRI. Those men with persistent highly suspicious lesions will under MRFTB. The biopsy results will be compared with intensity of Axumin uptake within the prostate. The urologist will have the discretion to biopsy Axumin avid lesions not detected by MRI.

ELIGIBILITY:
Inclusion Criteria:

* The participant has undergone MRFTB of an MRI lesion at the Department of Urology or at NYU Langone Health within past 12 months and has signed informed consent to participate in the NYU Urology prostate biopsy database.
* The most recent MRFTB of a PIRADS 4 or 5 lesion did not show clinically significant prostate cancer.

Exclusion Criteria:

* The urologist who performed the initial MRFTB does not feel a repeat MRI is indicated.
* Any contraindication to prostate biopsy including untreated urinary tract infection
* Prior allergic reaction to axumin
* Patient refuses MRI

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with negative prostate biopsy | 12 Months
  This will be measured by determining is if PET imaging with 18-F fluciclovine (Axumin) identifies those men with prior negative MRFTBs of PI-RADS 4 and 5 lesions who harbor clinically significant prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lepor, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The objective of the study is: to determine if PET imaging with 18-F fluciclovine identifies those men with prior negative MRFTBs of PI-RADS 4&5